CLINICAL TRIAL: NCT01448889
Title: Normobaric Hyperoxygenation for Prevention of Contrast Induced Nephropathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Fany Tusia, medical center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: cino2
Record Dates: First submitted 2011-04-06; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Nephropathy
Keywords: contrast induced nephropathy; oxigen; coronary angiography
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100% oxigen (Active Comparator): patients will recive 100% oxigen in a mask with reservoir from the begginind of the procedure to 4 hours after its termination
  Interventions: Drug: 100% oxigen
- placebo (Placebo Comparator): patients will recive 21% oxigen (room air) in a mask with reservoir from the begginind of the procedure to 4 hours after its termination
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 100% oxigen — patients will recive 100% oxigen in a mask with reservoir from the begginind of the procedure to 4 hours after its termination
  Arms: 100% oxigen
Drug: placebo — patients will recive 21% oxigen (room air) in a mask with reservoir from the begginind of the procedure to 4 hours after its termination
  Arms: placebo

SUMMARY:
Acute renal failure induced by radiographic contrast agents is a known complication of coronary angiography.hypoxia plays a major role in the pathogenesis of Contrast induced nephropathy.

The aim of the current study is to investigate the effect of normobaric hyperoxygenation therapy on renal functions in patients at high risk for CIN undergoing coronary angiography.

The study is aimed to include 180 consecutive patients with estimated GFR base on the MDRD equation of less than 60 mL/min/1.73 m2 that are candidates for elective coronary angiography. Patients with acute renal failure, acute myocardial infarction, noncompensated congestive heart failure, hemodynamic instability, known sensitivity to contrast media and patients who had been exposed to contrast media during the last 3 months will be excluded. Patients with oxygen blood saturation of less than 94% at room air will also be excluded from the study.

Study protocol Patients will be randomly assigned to receive either 100% oxygen by mask (treated group) or breath room air (control group) for duration of 4 hours starting at the beginning of the angiographic procedure.

All patients will be treated with 0.9% salin and NAC. Coronary angiography will be performed using nonionic, low osmolar iodine (Ultravist®-370) (Schering, Berlin, Germany).

All patients will be hospitalized 1 day before and at least 24 hours following angiography. Blood samples for urea, creatinine and cystatin- C will be drawn on admission, 6, 24 and 48 hours after coronary angiography. Urine sample will be taken 24 hours before angiography and 6, 24 and 48 hours post angiography. In those urine samples the ratio between creatinine to Isoprostanes and NO will be evaluated.

DETAILED DESCRIPTION:
Acute renal failure induced by radiographic contrast agents is a known complication of coronary angiography. It has been demonstrated that following contrast media application the renal outer medullar blood flow is reduced, resulting in medullar ischemia. N-acetylcysteine (NAC) together with well hydration stands in the center of treatments to prevent contrast induced nephropaathy (CIN).

Since, hypoxia plays a major role in the pathogenesis of CIN it seems rational that further increase oxygen delivery to the renal tissue will further ameliorate the expected CIN.

The aim of the current study is to investigate the effect of normobaric hyperoxygenation therapy on renal functions in patients at high risk for CIN undergoing coronary angiography.

The study protocol was approved by the local Ethics Committee and each patient will give written informed consent before including in the study. The study is aimed to include 180 consecutive patients with estimated GFR base on the MDRD equation of less than 60 mL/min/1.73 m2 that are candidates for elective coronary angiography. Patients with acute renal failure, acute myocardial infarction, noncompensated congestive heart failure, hemodynamic instability, known sensitivity to contrast media and patients who had been exposed to contrast media during the last 3 months will be excluded. Patients with oxygen blood saturation of less than 94% at room air will also be excluded from the study.

Study protocol Patients will be randomly assigned to receive either 100% oxygen by mask (treated group) or breath room air (control group) for duration of 4 hours starting at the beginning of the angiographic procedure.

All patients will be treated with 0.9% salin and NAC. Saline o.9% hydration will be infused at a rate of 1 mL/kg/hour 12 hours before and 12 hours after coronary angiography. NAC 1g [Mucomyst 20% solution (Bristol-Meyers, New York, NY, USA)] will be administered orally twice daily 24 hours before and 24 hours after coronary angiography. Coronary angiography will be performed using nonionic, low osmolar iodine (Ultravist®-370) (Schering, Berlin, Germany).

All patients will be hospitalized 1 day before and at least 24 hours following angiography. Blood samples for urea, creatinine and cystatin- C will be drawn on admission, 6, 24 and 48 hours after coronary angiography. Urine sample will be taken 24 hours before angiography and 6, 24 and 48 hours post angiography. In those urine samples the ratio between creatinine to Isoprostanes and NO will be evaluated.

Laboratory analysis Two 10mL aliquots from each urine collection will be separated and stored at -70°C until analyzed for nitric oxide metabolites and urinary isoprostanes.

Measurement of urinary nitric oxide metabolites Metabolites of nitric oxide (NOx) (NO2+ NO3) will be measured in the urine samples. Total NO synthesis will be evaluated in duplicates, by a specific two-step photocolorimetric assay (R&D Systems, USA) by a protocol supplied by a manufacturer. The intensity of the developing color was measured in ELISA reader, at 540 nm wavelength.

Oxidative stress Oxidative stress will be assessed by measurement of urinary isoprostanes, which are secondary end products of lipid peroxidation and are known to be an accurate and sensitive marker of renal oxidative stress in vivo. STAT-8 isoprostane PGF2 content will be estimated by a specific EIA (Cayman Chemical Co., Ann Arbor, Mich., USA) based on a competition between 8-isoprostane and 8-isoprostane-alkaline phosphatase conjugate for a limited number of the specific STAT-8 isoprostane PGF2 antibody binding sites and subsequent reaction of the immobilized complex with p-nitrophenyl-phosphate. The intensity of the developing yellow color will be measured in ELISA reader at 405 nm wavelength.

Investigators involved in the measurement of blood urea, creatinin and cystatin-C and in the urinary NOx and isoprostanes will be blinded to the patients' treatment.

Statistical analysis The calculation of the sample size is based on the following assumption: Baseline frequency of CIN of 20%, at least 35% reduction in the control group, alpha error level of 5%, beta error level of 50% and expected drop out rate of 15%.

Continuous baseline variables will be compared between the treatment groups by an unpaired t test and by a paired t test within each group. Categorical parameters will compared by a chi-square test. The effect of oxygen therapy on serum urea, creatinine, serum urea, serum cystatin-C, urinary NOx, and urinary isoprostanes at baseline 6, 24 and 48 hours following angiography will be compared between the groups by a general linear model repeated-measures analysis of variance (ANOVA). The statistical software SPSS (version 13.0, SPSS, Inc., Chicago, IL, USA) will be used for all analyses. All tests were two tailed. P values below 0.05 were considered significant. Data are expressed as mean SEM.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary angiography
* estimated GFR base on the MDRD equation of less than 60 mL/min/1.73 m2
* inform consent

Exclusion Criteria:

* acute renal failure
* acute myocardial infarction
* noncompensated congestive heart failure
* hemodynamic instability
* known sensitivity to contrast media
* patients who had been exposed to contrast media during the last 3 months
* Patients with oxygen blood saturation of less than 94% at room air.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
contrast induced nephropathy | 48 hours

SECONDARY OUTCOMES:
Nitric Oxide in urine sample | day -1, and 6,24,48 hours after exposure
urinary isoprostanes | day -1, and 6,24,48 hours after exposure
blood urea and creatinin | day -1, and 6,24,48 hours after exposure
cystatin-C | day -1, and 6,24,48 hours after exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Cardiac Care Unit, assaf harofhe medical center, Ẕerifin, Israel